CLINICAL TRIAL: NCT05726955
Title: The Effect of Exercise Applied With Stretching Platform on Pain, Proprioception, Balance, and Mobility in Patients With Chronic Low Back Pain
Brief Title: The Effect of Exercise Applied With Stretching Platform in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FU
Record Dates: First submitted 2023-01-13; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; exercise; balance; proprioception; mobility
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Masking Description: The evaluations of pain, proprioception, mobility, balance, functionality and quality of life were performed by a physiotherapist, while treatment programs were performed by the other physiotherapist in this study. Physiotherapists were blind to each other. Face to face interview method was used for the data collection. A consultation was provided by the researchers when the patients had questions. It took about 30 min to complete all assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control
- Exercise (Experimental): Group 2 (n=28) were included in an exercise training program applied with conservative treatment and a stretching platform (ETSP)
  Interventions: Other: Exercise training program

INTERVENTIONS:
Other: Exercise training program — an exercise training program applied with conservative treatment and a stretching platform (ETSP) 3 days a week for 6 weeks
  Arms: Exercise

SUMMARY:
This study aimed to examine and compare the effects of exercises applied with a stretching platform in addition to conservative treatment and conservative treatment only on pain, proprioception, balance, and mobility in patients with chronic low back pain. 55 people with chronic low back pain were included in the study and randomly divided into 2 groups. The participants in group 1 were included in the conservative treatment program, while the participants in group 2 were included in the exercise program applied with a stretching platform in addition to the conservative treatment. Pain intensity with Visual Analog Scale (VAS), proprioception sense with the active re-creation of passive positioning method without extremity support, mobility with Modified Schober Test (MST), Hand Finger-Ground Distance Measurement and Trunk Lateral Bending Measurement, balance level with Functional Reach Test, functionality with Oswestry Disability Index and quality of life was assessed with the EuroQol Group 5D-3L Questionnaire.

In the study, statistically significant differences were observed between the results of pain, proprioception, MST, HFGDM and TLBM, FRT, ODI and EuroQol Group 5D-3L in intragroup evaluations (p<0,05). In intergroup analysis, the VAS score during activity and 15° right ankle plantar flexion in proprioception evaluation were superior in the Group 2 compared to the group 1 (p<0.05).

It was observed that CT and exercises applied with a stretching platform in the treatment of chronic low back pain had positive effects on pain, proprioception, mobility, balance, functionality, and quality of life.

DETAILED DESCRIPTION:
Our study, which was designed as a randomized controlled prospective clinical trial, was conducted in accordance with the Declaration of Helsinki. Ethics committee approval for this study was obtained from University Ethics Committee with decision number (Study protocol: 6). The study included 55 participants aged 25-65 years, who had LBP for more than 12 weeks and whose pain intensity was greater than 3 on the 10 cm Visual Analog Scale (VAS). Those who have structural deformity, circulatory disorder, and a disease that will prevent mobility in the columna vertebralis, those who have undergone surgery for the columna vertebralis and lower extremity in the last year, and those diagnosed with vertigo and osteoporosis were not included in the study. All volunteers participating in the study were given an Informed Volunteer Consent Form and their signed consent was obtained.

2.2. Randomization The participants were randomized via the "Research Randomiser" website10. The numbers obtained as a result of randomization by entering the number of participants (n=55) and the number of groups (Group 1 and Group 2) were put into envelopes. Participants were assigned to groups according to the numbers on the envelopes they drew. Randomization was done in secret, blinding the groups and preventing the participants from meeting with the other group.

2.3. Groups Group 1 (n=27) were included in a conservative treatment program (CT) and the Group 2 (n=28) were included in an exercise training program applied with conservative treatment and a stretching platform (ETSP) 3 days a week for 6 weeks. Severity of pain, proprioception, mobility, balance, functionality, and quality of life (QoL) assessments of all participants were performed before and after the treatment. .

2.4. Assessments Demographic data including age, height, body weight, body mass index (BMI), previous diseases, and smoking habits of the participants who participated in the study were evaluated.

To evaluate the severity of pain, at night, at rest, and during activity, the VAS was used, which digitizes the parameter values that cannot be measured numerically, by numbering them from 0 to 10, where "0" is no pain and "10" is very severe pain11.

In the method of actively recreating passive positioning without supporting the extremity, in which a goniometer is used to evaluate the proprioception sense, the extremity was passively moved to the target angle while the participant's eyes were closed, and the participant returned to the starting point after focusing on the position for 10 seconds. The participant tried to find the target angle by actively moving the same extremity, and the difference was recorded as the deviation angle12.

Modified Schober Test (MST), Hand Finger-Ground Distance Measurement (HFGDM), and Trunk Lateral Bending Measurement (TLBM) were used to evaluate the level of mobility. In the MST, 5 cm below and 10 cm above the line connecting the spinal iliaca posterior superior were marked with the help of a tape measure while the participant was in an upright position. While the participant was performing maximum trunk flexion, the distance between the two points was measured and 15 cm was subtracted from this measurement. If the difference is less than 5 cm, it is MST (+). This result indicates that lumbar region mobility decreases13-14. In HFGDM, the participant is asked to bend forward and perform maximum flexion while in an upright position. In TLBM, the participant was asked to lean to the side with his arms on both sides of the body, with his shoulder and gluteal region resting against the wall. In both measurements, the distance between the third finger and the ground was measured with the help of a tape measure. Lumbar mobility increases as the distance between the finger and the floor decrease in TLBM and HFGDM15.

Functional Reach Test (FRT) was used for balance assessment. The participant was positioned to stand sideways against the wall. The shoulder on the wall was brought to 90° flexion and the elbow to full extension, and the participant was asked to make a fist with the same arm. The alignment of the 3rd metacarpal head was marked on the wall. The participant reached forward with the knees fully extended and the level of the 3rd metacarpal head was marked again. The difference between the two marks was measured with a tape measure. The average value was obtained after 3 trials. The same application was repeated with the eyes closed. The greater the difference between the marked points in FRT, the better the balance16-17.

The Oswestry Disability Index (ODI) was used for functionality assessment. ODI is a scale that evaluates the degree of loss of function in low back pain between "0" and "100" points. As the score in ODI increases, the level of disability increases18.

The EuroQol Group 5-Dimension 3-Level (EQ-5D-3L) QoL Scale was used for QoL assessment. The 1st item of the parameters evaluated in the 1st part of the scale includes the expressions "no problem", the 2nd item "moderately severe problem" and the 3rd item "very severe problem". In scoring, '11111' represents complete well-being, and '33333' represents coma or death. Section 2 contains VAS, with 100 representing "excellent health" and 0 for "very poor health"19-20.

2.5. Treatment Program All participants included in the study received conservative treatment, 3 days a week for 6 weeks. Conservative treatment included a 20-minute hot pack and conventional Transcutaneous Electrical Nerve Stimulation (TENS) and William's flexion exercises applied to the lumbar region. The exercises performed on the stretching platform designed to stretch the lumbar, gluteal, and posterior parts of the lower extremity were applied only to the participants in Group 2 for 3 days a week for 6 weeks after Williams flexion exercises.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 25-65 years,
* who had LBP for more than 12 weeks
* whose pain intensity was greater than 3 on the 10 cm Visual Analog Scale (VAS).

Exclusion Criteria:

* have structural deformity, circulatory disorder,
* have a disease that will prevent mobility in the columna vertebralis,
* those who have undergone surgery for the columna vertebralis and lower extremity in the last year,
* those diagnosed with vertigo and osteoporosis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 months
  To evaluate the severity of pain, at night, at rest, and during activity, the VAS was used, which digitizes the parameter values that cannot be measured numerically, by numbering them from 0 to 10, where "0" is no pain and "10" is very severe pain.

SECONDARY OUTCOMES:
measurement of proprioception sense, the method of actively recreating passive positioning without supporting the extremity | 6 months
  In the method of actively recreating passive positioning without supporting the extremity, in which a goniometer is used to evaluate the proprioception sense, the extremity was passively moved to the target angle while the participant's eyes were closed, and the participant returned to the starting point after focusing on the position for 10 seconds. The participant tried to find the target angle by actively moving the same extremity, and the difference was recorded as the deviation angle.
Modified Schober Test | 6 months
  assessment of mobility, the MST, 5 cm below and 10 cm above the line connecting the spinal iliaca posterior superior were marked with the help of a tape measure while the participant was in an upright position. While the participant was performing maximum trunk flexion, the distance between the two points was measured and 15 cm was subtracted from this measurement. If the difference is less than 5 cm, it is MST (+). This result indicates that lumbar region mobility decreases.
Functional Reach Test (FRT) | 6 months
  assessment of balance
The Oswestry Disability Index (ODI) | 6 months
  assessment of functionality
The EuroQol Group 5-Dimension 3-Level (EQ-5D-3L) | 6 months
  assessment of quality of life
Hand Finger-Ground Distance Measurement | 6 months
  In HFGDM, the participant is asked to bend forward and perform maximum flexion while in an upright position.In both measurements, the distance between the third finger and the ground was measured with the help of a tape measure. Lumbar mobility increases as the distance between the finger and the floor decrease in HFGDM.
Trunk Lateral Bending Measurement | 6 months
  In TLBM, the participant was asked to lean to the side with his arms on both sides of the body, with his shoulder and gluteal region resting against the wall. In both measurements, the distance between the third finger and the ground was measured with the help of a tape measure. Lumbar mobility increases as the distance between the finger and the floor decrease in TLBM.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydin, PhD, Principal Investigator — Firat University
Locations (1):
- Fizyopedi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammad NS, Nazli R, Zafar H, Fatima S. Effects of lipid based Multiple Micronutrients Supplement on the birth outcome of underweight pre-eclamptic women: A randomized clinical trial. Pak J Med Sci. 2022 Jan-Feb;38(1):219-226. doi: 10.12669/pjms.38.1.4396. PMID 35035429